CLINICAL TRIAL: NCT02454205
Title: Evaluating a New Treatment Regimen for Patients With Multidrug-resistant TB (MDR-TB) - a Prospective Open-label Randomised Controlled Trial
Brief Title: An Open-label RCT to Evaluate a New Treatment Regimen for Patients With Multi-drug Resistant Tuberculosis
Acronym: NEXT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Limpopo (Other); Walter Sisulu University (Other); University of Stellenbosch (Other); University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Principle Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NExT-5001
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Tuberculosis; Multidrug Resistant Tuberculosis; Extensively-drug Resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — Linezolid; bedaquiline; Levofloxacin; Pyrazinamide; Isoniazid; Ethionamide; terizidone; Moxifloxacin; Kanamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment 21-24 months (Active Comparator): Participants will receive a 6-8 month intensive phase of: Kanamycin IM 500-750mg (40-50kg) or 1000mg (51-90kg) daily, Moxifloxacin 400mg od, Pyrazinamide 1000-1750mg (40-50kg) or 1750-2000mg (51-70kg) or 2000-2500mg (71-90kg) daily, Ethionamide 500mg (40-50kg) or 750mg (51-70kg) or 750-1000mg (71-90kg) daily,Terizidone 750mg (40-70kg) or 750-1000mg (71-90kg) daily.
  The continuation phase will start after 2 consecutive negative sputum cultures and continue for 18 months with Moxifloxacin, PZA, Ethionamide and Terizidone.
  In 2016 the WHO revised the treatment guidelines for MDR-TB. The South African National Tuberculosis Program adopted these recommendations and it was integrated into the study in September 2016: SA NTP recommended shorter regimen(9-12 months):Intensive phase (4-6 months): kanamycin, levofloxacin, clofazimine, pyrazinamide, high-dose isoniazid/ethionamide, ethambutol. Continuation phase (5 months): levofloxacin, clofazimine, pyrazinamide, ethambutol.
  Interventions: Drug: Pyrazinamide; Drug: Ethionamide; Drug: Terizidone; Drug: Moxifloxacin; Drug: Kanamycin
- Interventional treatment 6-9 months (Experimental): Participants will receive six to nine months of oral:
  Linezolid 600mg daily (reduce to 300mg if toxicity occurs), Bedaquiline 400mg for 2 weeks, followed by 200mg three times per week, Levofloxacin 750mg (<50kg) or 1000mg (>50kg) daily, PZA 1000-1750mg (40-50kg) or 1750-2000mg (51-70kg) or 2000-2500mg (71-90kg) daily, Ethionamide 15mg/kg (max 900mg) daily, or high-dose Isoniazid 500mg (40-50kg) or 750mg (51-70kg) or 750-1000mg (71-90kg) daily, or Terizidone 750mg (40-70kg) or 750-1000mg (71-90kg) daily.
  A gene-directed diagnostic approach will be used in the interventional arm to individualise therapy and to inform on the use of high dose INH versus ethionamide. Treatment will stop after 3 consecutive negative sputum cultures.
  Interventions: Drug: Linezolid; Drug: Bedaquiline; Drug: Levofloxacin; Drug: Pyrazinamide; Drug: Isoniazid; Drug: Ethionamide; Drug: Terizidone

INTERVENTIONS:
Drug: Linezolid — 600mg Linezolid po daily, reduced to 300mg po daily if toxicity occurs.
  Arms: Interventional treatment 6-9 months
Drug: Bedaquiline — 400mg po daily for 2 weeks, followed by 200mg three times per week .
  Arms: Interventional treatment 6-9 months
Drug: Levofloxacin — 750mg (<50kg) 1000mg (>50kg)
  Arms: Interventional treatment 6-9 months
Drug: Pyrazinamide — 1000-1750mg (40-50kg) 1750-2000mg (51-70kg) 2000-2500mg (71-90kg)
  Other Names: PZA
Drug: Isoniazid — high dose Isoniazid 500mg (40-50kg) 750mg (51-70kg) 750-1000mg (71-90kg)
  Other Names: INH
  Arms: Interventional treatment 6-9 months
Drug: Ethionamide — 15mg/kg (max 900mg)
Drug: Terizidone — 750mg (40-70kg) 750-1000mg (71-90kg)
Drug: Moxifloxacin — 400mg po daily.
  Arms: Conventional treatment 21-24 months
Drug: Kanamycin — 500-750mg (40-50kg) 1000mg (51-90kg) intramuscular daily during 6-8 month intensive phase.
  Arms: Conventional treatment 21-24 months

SUMMARY:
This study aims to evaluate the impact of a new injection-free six-to-nine month treatment regimen of linezolid, bedaquiline, levofloxacin, pyrazinamide (PZA) and ethionamide/high dose isoniazid (INH) compared to the conventional empiric injection-based regimen. The secondary aim is to determine if other treatment-related outcomes including adverse events, adherence to treatment, culture conversion, and cure/completion are significantly different in the intervention and conventional arms.

DETAILED DESCRIPTION:
Background:

TB is completely out of control in South Africa and is now officially the most common cause of death in this country. Alarmingly, the gravity if this pandemic has now been compounded by the emergence of multidrug-resistant TB (MDR-TB), which constitutes resistance to the two most potent anti-tuberculous drugs, namely rifampicin and isoniazid . XDR-TB refers to resistance to rifampicin, isoniazid, any fluoroquinolone, and any second line injectable drug (amikacin, kanamycin, or capreomycin). MDR-TB is a burgeoning epidemic in South Africa, with rates trebling over the last decade. It is of considerable concern because mortality is high (up to 50% in South Africa) and it often affects economically active young adults. It is also a major threat to health care workers in South Africa. We recently showed a rate in SA health care workers 6 fold higher than the general population further exacerbating the shortage of this critical workforce in the country. The increasing cost to manage this disease is unsustainable.

Although drug-resistant TB comprises less than 2% of the total caseload in the country (approximately ½ million patients with TB treated per year), it consumes almost 40% of the total national TB programme budget, and more than 60% of the total TB drug budget. This is not sustainable and drug-resistant TB therefore has the capacity to destabilise functional TB control programmes in many countries in Africa.

The treatment of MDR-TB is arduous, with a six to eight month intensive phase of daily painful injections of Kanamycin combined with oral pyrazinamide, a fluoroquinolone (moxifloxacin or levofloxacin), prothionamide and either cycloserine or para-aminosalicylic acid (if cycloserine cannot be used). Treatment continues for 18 months after consecutive negative sputum cultures, and lasts at least 20 months. There are substantial drug-associated toxicities and adverse events that frequently lead to interruption or cessation of treatment.

This study proposes to test the efficacy of a new drug regimen for the treatment of MDR-TB which is of short term duration and which does not contain an injectable drug, thus making treatment easier to administer and thereby potentially increasing compliance. All the drugs will be available to the NTP if the study is shown to be successful. This regimen will comprise linezolid, bedaquiline, levofloxacin, PZA and either ethionamide or high dose INH or teridazone. A gene-directed diagnostic approach (mutational analysis) will be used in the interventional arm to individualise therapy and to inform on the use of high dose INH versus ethionamide. If both mutations are present then to administer teridazone.

Furthermore, in the proposed study the key aim is to test a regimen (rather than an individual drug) and will look at how the outcomes (24 month), including treatment completion/cure (i.e. treatment success which is the primary outcome) and mortality, are impacted. It is expected that introduction of a shortened effective regimen will reduce drop out and drastically reduce mortality and on-going transmission. Moreover, the rates of XDR-TB and TDR-TB may also decline.

The study will be conducted at 5 trial sites in South Africa that are designated MDR-TB treatment facilities and it many cases patients will be recruited from the satellite clinics of these centres reflecting the decentralized MDR-TB program. All the sites have the necessary expertise and facilities to carry out the proposed study. The study is a fully conceived and funded within South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed culture and/or GeneXpert positive pulmonary TB.
* Rifampicin resistance detected using at least two susceptibility testing assays (GeneXpert, HainMTBDRplus or phenotypic) using a sputum sample during screening.
* Provide written informed consent prior to all trial-related procedures including HIV testing.
* Male or female aged 18 years and older.
* Body weight between 40 and 90 kg, inclusive.
* Women of non-childbearing potential or participants of either sex who are using or willing to use effective methods of birth control

Exclusion Criteria:

* A participant who in the opinion of the investigator is unlikely to cope with regular visits to the trial site either because of travel constraints, or because of drug or alcohol abuse, or other reason.
* Known at screening to have XDR-TB or pre-XDR-TB (i.e. fluoroquinolone or second-line injectable drug (SLID) resistance i.e. to capreomycin, amikacin and kanamycin).
* Previous history of treatment for MDR-TB or XDR-TB or previous treatment with bedaquiline.
* Currently on MDR-TB treatment for more than 2 weeks.
* Any participant with a Karnofsky score < 50.
* Known allergy to any of the trial drugs or related substances.
* Having participated in other clinical studies within 8 weeks prior to trial start where investigational agents were used that may potentially impact current trial outcome.
* Presence (or evidence) of symptomatic neuropathy grade 3 or higher.
* Epilepsy where drugs prolonging QT interval are used.
* Participant who is pregnant, breast-feeding (and not willing to stop), or planning to conceive a child within 6 months of cessation of treatment.
* Incompatibility between microbiological and clinical/ radiological findings (i.e. where the clinical and/or radiological findings are discordant with microbiological testing suggesting laboratory contamination).
* Participants with ECG abnormalities, in particular QT prolongation.
* Any pre-existing laboratory abnormality which in the opinion of the investigator will place the participant at risk. Patients with any of the following baseline laboratory abnormalities will be excluded from the study:

  * Creatinine grade 2 or worse (>1.4 times ULN)
  * Hemoglobin level grade 4 (HB <6.5g/dL)
  * Platelets grade 3 or worse (<49999 x 109/L)
  * ALT grade 3 or worse (>5 times ULN)
  * Total bilirubin grade 3 or worse (>2.5 times ULN)
* Specific prior or concurrent medication/treatments (see Restrictions section below, Table 3).
* Rifampicin monoresistant TB.
* Fluoroquinolone and/or SLID resistance. Although in South Africa, the standard of care does not single out MDR-TB with fluoroquinolone or aminoglycoside resistance at initiation of MDR-TB treatment, in this study the Hain MTBDRsl LPA will be used on the sputum sample to exclude any pre-XDR and XDR cases from participation in the study (results from the LPA and phenotypic DST testing on the isolate will be available 3-6 weeks later).

All inclusion and no exclusion criteria must be met prior to enrolment and randomisation. Whenever the investigator has reason to suspect that there might be a health problem (other than TB) participation should only be considered after discussing the case with the medical monitor. Note: Participants who are currently on, or have previously been on drug-sensitive TB treatment are not excluded from participation.

Post-randomisation exclusion criteria:

• Fluoroquinolone and/or SLID resistance detected on DST using the isolate. Note: A woman who falls pregnant during the treatment phase of the trial will not be excluded but will be counselled regarding potential termination of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Treatment success | 24 months after initiation of treatment in either arm.
  In the conventional arm treatment success is defined as the sum of cured or treatment completed cases. In the intervention arm treatment success is defined as the sum of cured and treatment completed cases, without subsequent relapse, re-infection or death during the 15-18 month follow up period.

SECONDARY OUTCOMES:
Favourable outcome rate | At 6-9 months for the intervention arm and 21-24 months for the conventional arm.
Time specific rate of treatment failure. | 6-36 months
Time specific culture conversion proportions and rates. | 6-36 months
Time specific relapse rate. | 6-36 months.
Rate of re-infection. | 6-36 months.
All cause mortality | 0-36 months.
Composite measure of QT interval on ECG, grade 3 and 4 adverse events, stopping drugs Safety and tolerability end-points. | 0-36 months.
Default rate | 2-24 months
  Rate at which participants interrupt treatment for two or more consecutive months for any reason without medical approval.
Rate of loss of follow-up. | 0-36 months.
  Rate at which a participant becomes untraceable at any point in the study, and remains untraceable at completion of study despite every effort being made by researchers to locate the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MBChB, Principal Investigator — UCT Lung Institute
Locations (1):
- Brooklyn Chest Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esmail A, Oelofse S, Lombard C, Perumal R, Mbuthini L, Goolam Mahomed A, Variava E, Black J, Oluboyo P, Gwentshu N, Ngam E, Ackerman T, Marais L, Mottay L, Meier S, Pooran A, Tomasicchio M, Te Riele J, Derendinger B, Ndjeka N, Maartens G, Warren R, Martinson N, Dheda K. An All-Oral 6-Month Regimen for Multidrug-Resistant Tuberculosis: A Multicenter, Randomized Controlled Clinical Trial (the NExT Study). Am J Respir Crit Care Med. 2022 May 15;205(10):1214-1227. doi: 10.1164/rccm.202107-1779OC. PMID 35175905
- [Derived] Wasserman S, Huo S, Ky K, Malig YN, Esmail A, Dheda K, Bacchetti P, Gerona R, Maartens G, Gandhi M, Metcalfe J. Correlation of Linezolid Hair Concentrations with Plasma Exposure in Patients with Drug-Resistant Tuberculosis. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e02145-19. doi: 10.1128/AAC.02145-19. Print 2020 Feb 21. No abstract available. PMID 31932382
- See also: Home page of the Lung Institute — http://www.lunginstitute.co.za